CLINICAL TRIAL: NCT04918004
Title: The Effect of Sleep hygıene traınıng gıven to patıents wıth dıabetes mellıtus on Blood Sugar regulatıon: a randomızed Controlled Study
Brief Title: The Effect of Sleep hygıene traınıng on Blood Sugar regulatıon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Süleyman Görpelioğlu, Clinical Professor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 27.11.2017 - 43/06
Record Dates: First submitted 2021-05-30; First posted 2021-06-08 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2; Sleep Hygiene
Keywords: Diabetes Mellitus Type 2; Sleep Hygiene; Treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): Patients in the case group were given one-to-one sleep hygiene training by researchers and, a brochure containing 10 lifestyle changes related to sleep hygiene as well as they assessed at the first interview and the last interview, received routine health care, and
  Interventions: Behavioral: Sleep Hygiene
- Control group (No Intervention): Patients in the control group were assessed at the first interview and the last interview, received routine health care, and no intervention was performed during the research.

INTERVENTIONS:
Behavioral: Sleep Hygiene — 1. One-to-one sleep hygiene training, the content of which was created by the researchers,
  2. A brochure containing 10 lifestyle changes related to sleep hygiene
  Arms: Case group

SUMMARY:
Although many studies have shown an inverse relationship between blood glucose regulation and sleep hygiene, recommendations for improving sleep hygiene have not yet been included in diabetes treatment guidelines. In this study, it was aimed to reveal with a randomized controlled study whether training on sleep hygiene will have an effect on blood glucose regulation of Type 2 diabetes patients. Case and control groups will be formed by random sampling method. Pıttsburgh sleep quality index will be applied face to face and HbA1c values will be recorded for all patients included in the study. In addition, sleep hygiene training will be given to the case group. Among the patients included in the study, the second HbA1c levels of those who came for routine diabetes control within six months will be recorded and the sleep hygiene education compliance scale will be applied to the case group. Differences between groups will be evaluated using chi-square and Student's t tests. According to the results of the research, it will be tried to decide whether sleep hygiene education can be used in the treatment of type 2 diabetes patients.

DETAILED DESCRIPTION:
Although there are many studies in the literature examining the relationship between diabetes mellitus and poor sleep quality, most of the studies are cross-sectional. While the relationship between sleep quality and blood glucose regulation was clearly shown in these studies, very few studies aimed to observe the effect of sleep quality correction on blood glucose regulation. As a result of this, of the 35 guidelines addressed in a meta-analysis conducted in 2020 only 14 guidelines included sleep in their recommendations, optimising sleep duration and quality and the management of sleep disorders were discussed as a therapeutic approach in 6 guidelines. In these also only 3 guidelines recommended optimal sleep duration as a therapeutic target of life style intervention and self-management education with one guideline identifying optimal sleep as a means of achieving glycaemic targets in T2DM .

In this randomised controlled study, it is aimed to provide evidence for the guidelines on the treatment of diabetes by demonstrating whether the education that includes simple lifestyle changes to increase sleep hygiene will have an effect on blood glucose regulation of Type 2 diabetes patients.

In the power analysis based on the tests to be used, when Type 1 error (α) = 0.05, Type 2 error (1-β) = 0.95, effect size is considered as 0.5; it was calculated that the sample size should be 210 (105 for each group) in total.

Patients with sleep disorders, language or psychiatric problems known to interfere with responding to the questionnaire, and patients whose antidiabetic treatment was changed at the first control examination will be excluded from the study.

In their first visit, the participants will be administered a routine diabetes control including HbA1c measurements, as well as a sociodemographic data collection questionnaire prepared by the researchers, a questionnaire consisting of 20 questions including questions about diabetes and sleep problems, and the Turkish version of the Pittsburgh Sleep Quality Index (PSQI) by face-to-face interview technique.

In addition, each patient included in the case group was given a brochure containing one-on-one sleep hygiene education and 10 lifestyle changes related to sleep hygiene, the content of which was created by the researchers.

Recommendations in the sleep hygiene leaflet :

* Enter the bed when you feel sleepy. If you lie in bed for more than half an hour, get out of bed. When you feel sleepy, go back to bed
* Do not sleep more than 1 hour during the day time.
* Avoid heavy and fatty meals in the evening, do not go to bed very hungry or very satiated. Avoid beverages such as coffee, tea, coke, energy drinks and alcohol.
* Exercise or walk regularly in the evening, but avoid physically strenuous activities 3-4 hours before bedtime
* In order for your body clock to work properly, live regularly. Get out of bed at the same time everyday. Wake up at the time you should wakeup in the morning, even if you went to bed at a different time of the night. Follow this rule, even on the weekend, and make it a habit to always get up at the same time. Sleeping and awakening times are important in maintaining sleep patterns.
* Use the bed for sleep purposes only. Do not do activities such as eating, watching TV, reading a book, or planning the next day in bed.
* Make sure your bedroom is quiet and dark
* Avoid exciting activities such as watching horror movies or reading adventure boks before going to bed
* Try to avoid a stressful life.
* Never take sleeping pills without your doctor's knowledge.

At the next visit of all participants, a second visit PSQI will be administered in addition to HbA1c, and a statement-based "sleep hygiene education compliance questionnaire" will be administered to the case group, questioning whether they have complied with the items in the sleep hygiene education material recommended at the first interview.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were admitted to our clinic with the diagnosis of diabetes mellitus type 2 during the study

Exclusion Criteria:

* Patients with a known sleep disorder,
* Language or psychiatric problems that prevented responding to the questionnaire
* Patients who underwent changes in their antidiabetic treatment during the first control examination
* Those who did not re-admit to the hospital for routine check-ups within 6 months after the first visit
* Patients who declared not to comply with the recommendations were excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Pıttsburgh Sleep Quality Index Score | Within 3-6 months after first visit
  Pıttsburgh sleep quality index score was used in order to determine whether the training provided increases the sleep quality or not.An increase in the second measured index score compared to the first measured Pitssburg sleep quality index score will indicate a decrease in sleep quality.
Hba1c mmol/mol | Within 3-6 months after first visit
  To detect change in blood sugar regulation HbA1c values will be used. A decrease in the second measured HbA1c values compared to the first measured HbA1c values will indicate a positive effect on blood sugar regulation .

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Görpelioğlu, Prof.Dr., Principal Investigator — Academic staff
Locations (1):
- University of Health Sciences Turkey Ankara Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kachi Y, Nakao M, Takeuchi T, Yano E. Association between insomnia symptoms and hemoglobin A1c level in Japanese men. PLoS One. 2011;6(7):e21420. doi: 10.1371/journal.pone.0021420. Epub 2011 Jul 1. PMID 21747936
- [Background] Tan X, van Egmond L, Chapman CD, Cedernaes J, Benedict C. Aiding sleep in type 2 diabetes: therapeutic considerations. Lancet Diabetes Endocrinol. 2018 Jan;6(1):60-68. doi: 10.1016/S2213-8587(17)30233-4. Epub 2017 Aug 24. PMID 28844889
- [Background] Nedeltcheva AV, Scheer FA. Metabolic effects of sleep disruption, links to obesity and diabetes. Curr Opin Endocrinol Diabetes Obes. 2014 Aug;21(4):293-8. doi: 10.1097/MED.0000000000000082. PMID 24937041
- [Background] Spiegel K, Tasali E, Leproult R, Van Cauter E. Effects of poor and short sleep on glucose metabolism and obesity risk. Nat Rev Endocrinol. 2009 May;5(5):253-61. doi: 10.1038/nrendo.2009.23. PMID 19444258
- [Background] Lee SWH, Ng KY, Chin WK. The impact of sleep amount and sleep quality on glycemic control in type 2 diabetes: A systematic review and meta-analysis. Sleep Med Rev. 2017 Feb;31:91-101. doi: 10.1016/j.smrv.2016.02.001. Epub 2016 Feb 9. PMID 26944909
- [Background] Smyth A, Jenkins M, Dunham M, Kutzer Y, Taheri S, Whitehead L. Systematic review of clinical practice guidelines to identify recommendations for sleep in type 2 diabetes mellitus management. Diabetes Res Clin Pract. 2020 Dec;170:108532. doi: 10.1016/j.diabres.2020.108532. Epub 2020 Nov 4. PMID 33157114
- [Background] Zhu B, Hershberger PE, Kapella MC, Fritschi C. The relationship between sleep disturbance and glycaemic control in adults with type 2 diabetes: An integrative review. J Clin Nurs. 2017 Dec;26(23-24):4053-4064. doi: 10.1111/jocn.13899. Epub 2017 Jul 17. PMID 28544107
- [Background] Chasens ER, Korytkowski M, Sereika SM, Burke LE. Effect of poor sleep quality and excessive daytime sleepiness on factors associated with diabetes self-management. Diabetes Educ. 2013 Jan-Feb;39(1):74-82. doi: 10.1177/0145721712467683. Epub 2012 Nov 27. PMID 23192600
- [Background] Seibert PS, Valerio J, DeHaas C. The concomitant relationship shared by sleep disturbances and type 2 diabetes: developing telemedicine as a viable treatment option. J Diabetes Sci Technol. 2013 Nov 1;7(6):1607-15. doi: 10.1177/193229681300700621. PMID 24351187
- [Background] Larcher S, Benhamou PY, Pepin JL, Borel AL. Sleep habits and diabetes. Diabetes Metab. 2015 Sep;41(4):263-271. doi: 10.1016/j.diabet.2014.12.004. Epub 2015 Jan 23. PMID 25623152
- See also: TEMD Diabetes Mellitus Çalışma ve Eğitim Grubu, Diagnosis and Monitoring Guide for Diabetes Mellitus and Its Complications 2020 Türkiye Endokrinoloji ve Metabolizma Derneği: 2020. p.40-44 — https://temd.org.tr/admin/uploads/tbl_kilavuz/20200625154506-2020tbl_kilavuz86bf012d90.pdf
- See also: Agargün M Y, Kara H, Anlar O (1996) Validity and Reliability of Pittsburgh Sleep Quality. Türk Psikiyatri Dergisi, 7: 107-115. — http://www.turkpsikiyatri.com/default.aspx?modul=turkceOzet&gFPrkMakale=210
- See also: TurcosaAnalytics (2021). TURCOSA [Cloud-based statistical software]. — https://release.turcosa.com.tr/